CLINICAL TRIAL: NCT00783900
Title: Intravenous Metoprolol Versus Biatrial Pacing in the Prevention of Atrial Fibrillation After Cardiac Surgery
Brief Title: Intravenous Administration of Metoprolol Versus Biatrial Pacing in the Prevention of Atrial Fibrillation After Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: Oulu University Hospital (Other); Hospital Cordia, Kuopio, Finland (Unknown)
Responsible Party: Halonen Jari, Kuopio university hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KUH5204006; Eudra-CT: 2008-006932-36
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2011-11

CONDITIONS: Atrial Fibrillation; Biatrial Pacing; Metoprolol
Keywords: Prevention
MeSH Terms: conditions — Atrial Fibrillation | interventions — Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- metoprolol (Active Comparator)
  Interventions: Other: metoprolol, biatrial pacing
- biatrial pacing (Active Comparator)
  Interventions: Other: metoprolol, biatrial pacing

INTERVENTIONS:
Other: metoprolol, biatrial pacing — Prevention, atrial fibrillation, cardiac surgery, biatrial pacing, metoprolol

SUMMARY:
The aim of the study is to compare the effectiviness of biatrial pacing versus intravenous administration of metoprolol in the prevention of atrial fibrillation after cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* elective CABG and aortic valve cardiac patients,
* previous use of beta blocker

Exclusion Criteria:

* Previous episodes of Atrial fibrillation or flutter,
* II or II degree atrioventricular block, uncontrolled heart failure
* Sick sinus syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
biatriac pacing | 48 hours
Incidence of atrial fibrillation | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Halonen Jari, Kuopio, Finland